CLINICAL TRIAL: NCT01098591
Title: Meta-Analysis of Cell-based CaRdiac stUdiEs: ACCRUE
Acronym: ACCRUE
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Nantes University Hospital (Other); Oslo University Hospital (Other); Medical University of Silesia (Other); Hannover Medical School (Other); VZW Cardiovascular Research Center Aalst (Other); Cedars-Sinai Medical Center (Other); Johann Wolfgang Goethe University Hospital (Other); University of Ulm (Other); Military Medical Academy, Belgrade, Serbia (Other); Novosibirsk Scientific Research Institute for Circulatory Pathology (Other); Rigshospitalet, Denmark (Other); Asklepios Kliniken Hamburg GmbH (Other); Leiden University Medical Center (Other); University of Debrecen (Other); University of Targu Mures, Romania (Other); University Clinic for Cardiology, Skopje, Republic of Macedonia (Unknown); State Health Center, Hungary (Other); Karolinska Institutet (Other); University of Zurich (Other); University of Oulu (Other); Odense University Hospital (Other); Minneapolis Heart Institute (Other); The University of Texas Health Science Center, Houston (Other); Klinik Hirslanden, Zurich (Other); University Hospital, Toulouse (Other); Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Mariann Gyongyosi, MD PhD, Medical University of Vienna
Other Study IDs: MUW - Meta
Record Dates: First submitted 2010-03-30; First posted 2010-04-05 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Ischemic Heart Disease
Keywords: meta-analysis; stem cell; cardiac; remodeling; ACCRUE
MeSH Terms: conditions — Myocardial Ischemia | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Myocardial infarction: Patients with post-myocardial infarction receiving cell therapy either intracoronarily or intramyocardial
  Interventions: Other: cell therapy
- Ischemic cardiomyopathy: Patients with ischemic cardiomyopathy treated with cell therapy either intracoronarily or intramyocardial
  Interventions: Other: cell therapy

INTERVENTIONS:
Other: cell therapy

SUMMARY:
Numerous human cardiac stem cell studies have been published, including relatively small number of patients. Meta-analysis of randomized trials have reported safety and a 3-6% increase in global left ventricular performance after intracoronary stem cell therapy in patients with acute myocardial infarction. Since most of the studies used different type of stem cells, delivery modes, and patient population, the results are heterogenous, therefore the comparison of the results is biased regarding generalizable conclusions about the effect of treatment. The present comparative meta-analysis is based on individual patient data, and gathers and pools the raw data, and analyzes the clinical outcome, safety and efficacy of the cardiac stem cell therapy.

DETAILED DESCRIPTION:
* Background: Many clinical trials and meta-analyses presented moderate but significant improvement of the left ventricular ejection fraction (LVEF) after intracoronary autologous bone-marrow (BM) or peripheral blood origin stem cells transfer. However, it remains controversial, whether this beneficial effects is comparable with the intramyocardial delivery of the stem cells, or could be maintained during moderate and long term follow-up. The BOOST trial suggested that cardiac stem cell therapy did not improve LVEF at 5-year follow-up. By contrast, BALANCE study showed a long sustained benefit of BM-stem cells treatment. Due to these divergent outcomes of the presented trials, the aim of the present meta-analysis is to compare the safety and effectiveness of the cardiac stem cell therapy in different patient population, delivery mode and cell type, to find out, which patients with which therapy mode can have the greatest benefit from cardiac stem cell therapy.
* Study design: individual patient data meta-analysis
* Data sources: European Centre performing human cardiac stem cell therapy have been contacted calling for participation.
* Methods: Individual data gathering and entering into the database for a pooled analysis. The meta-analysis will be done in line with recommendation from the Cochrane Collaboration and the Quality of Reporting of Meta-analyses guidelines with Review Manager 5.0. Fixed-effect model will be used.

ELIGIBILITY:
Inclusion Criteria:

* patient included in one of the registered cell-based cardiac therapy of the participating center

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with cell-based cardiac therapy at one of the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Freedom from occurrence of major adverse cardiac and cerebrovascular events (MACCE), including all-cause death, re-infarction, revascularization and stroke | 12 months
  MACCE is defined as all-cause death, re-infarction, revascularization and stroke

SECONDARY OUTCOMES:
Hard clinical end point | 12 months
  all-cause death, re-infarction and stroke
Changes in end-diastolic volume | 12 months
  End-diastolic volume is an index of ventricular remodeling
Changes in end-systolic volume | 12 months
  Index of ventricular systolic performance
Changes in ejection fraction | 12 months
  Improvement of systolic cardiac function after cell therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mariann Gyongyosi, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Gyongyosi M, Wojakowski W, Lemarchand P, Lunde K, Tendera M, Bartunek J, Marban E, Assmus B, Henry TD, Traverse JH, Moye LA, Surder D, Corti R, Huikuri H, Miettinen J, Wohrle J, Obradovic S, Roncalli J, Malliaras K, Pokushalov E, Romanov A, Kastrup J, Bergmann MW, Atsma DE, Diederichsen A, Edes I, Benedek I, Benedek T, Pejkov H, Nyolczas N, Pavo N, Bergler-Klein J, Pavo IJ, Sylven C, Berti S, Navarese EP, Maurer G; ACCRUE Investigators. Meta-Analysis of Cell-based CaRdiac stUdiEs (ACCRUE) in patients with acute myocardial infarction based on individual patient data. Circ Res. 2015 Apr 10;116(8):1346-60. doi: 10.1161/CIRCRESAHA.116.304346. Epub 2015 Feb 19. PMID 25700037